CLINICAL TRIAL: NCT02374528
Title: Clinical Randomized Controlled Trials on Negative Pressure Wound Therapy for Skin Grafts
Brief Title: Negative Pressure Wound Therapy for Skin Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Jiayuan, Professor, vice director of surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015046
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Skin Transplantation
Keywords: Negative pressure wound therapy; wound; split-thickness skin grafting
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative pressure wound therapy (Experimental): Negative pressure wound therapy (NPWT) is the application of suction (negative pressure) to wounds with skin grafting.
  Interventions: Procedure: Negative pressure wound therapy
- standard pressure bolster dressing (Active Comparator): This method is traditional used in skin grafting wound.
  Interventions: Procedure: standard pressure bolster dressing

INTERVENTIONS:
Procedure: Negative pressure wound therapy — Negative pressure wound therapy (NPWT) is the application of suction (negative pressure) to wounds with skin grafting.
  Arms: Negative pressure wound therapy
Procedure: standard pressure bolster dressing — This method is traditional used in skin grafting wound.
  Arms: standard pressure bolster dressing

SUMMARY:
The repairing of various wounds is always a great challenge in burn surgery and plastic surgery. Skin-grafting is the main therapy. Bolster dressings are traditionally applied to secure the graft to the wound bed, however, there is some evidence to show that irregularly contoured recipient sites, poorly healing areas, reduce the success rate of skin-grafting with traditional bolster dressings, increasing morbidity, pain. Negative pressure wound therapy has been advocated as a potential solution to some of these issues. To further test the healing rate and safety of this new method, the investigators propose a prospective randomized controlled trial to compare this method with traditional bolster dressings application in skin-grafting.

DETAILED DESCRIPTION:
The repairing of various wounds is always a great challenge in burn surgery and plastic surgery. Skin-grafting is the main therapy. Bolster dressings are traditionally applied to secure the graft to the wound bed, however, there is some evidence to show that irregularly contoured recipient sites, exuding wounds, poorly healing areas, and the presence of shear stress significantly reduce the success rate of skin-grafting with traditional bolster dressings, increasing morbidity, pain, hospital stay, and cost. Negative pressure wound therapy (NPWT) has been advocated as a potential solution to some of these issues. the application of NPWT to skin-grafting may promote blood flow and microcirculation to the graft bed, reduction of edema, exudates, and hematomas, and result in significant qualitative improvement in split skin graft take. To further test the healing rate and safety of this new method, the investigators propose a prospective randomized controlled trial to compare this method with traditional bolster dressings application in skin-grafting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who need to skin graft to repair the wound
* Subjects signed the informed consent in the day of the age of not more than 85 years old (for minors, legal guardian should be signed)
* Stable vital signs, regular examination showed that subjects could tolerate surgery
* Subjects' mental state are good, could follow the doctor's advice, visit on a regular basis
* Understanding and willing to participate in this clinical trial and signed informed consent
* All women subjects must agree to take effective contraceptive measures in the six months study period, and without pregnancy before participate in the treatment
* No other serious diseases conflicts with the trail

Exclusion Criteria:

* Allergic constitution of negative pressure dressing
* Severe uncontrolled disease or acute systemic infections and complication with other serious heart, lung disease, encephalopathy and other organs or have a rapid progress or terminal disease
* Subjects with mental illness
* Subjects could not cooperate with the clinical trial personnel to finish trials
* Existing disease (malignant tumor, autoimmune disease) or require the use of drugs (high-dose glucocorticoids, which is defined as accepting 40 mg or more daily prednisone or prednisone amount, period of two weeks or more) will affect the healing of the wound
* For HIV positive patients, clinical diagnosis of patients with AIDS or the screening phase of neutrophil count (ANC) absolutely < 1000 cells/mm3
* Subjects could not tolerate surgery
* Subjects are unlikely to survive in the study period
* The investigators think that who should not be included
* Subjects are in or participated in other clinical researchers over the past 12 weeks
* Subjects are participated in this trial at any time in the past

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
healing rate (the percentage of subjects that achieved complete wound closure, complete wound closure is defined as skin complete reepithelialization without drainage or dressing requirements) | postsurgery week 4
  the percentage of subjects that achieved complete wound closure, complete wound closure is defined as skin complete reepithelialization without drainage or dressing requirements.

SECONDARY OUTCOMES:
VAS pain grade | postsurgery week 4
  assess the pain of the wound at each visit time
Skin graft survival rate | postsurgery week 2
  The area of the skin graft has been survival percentage accounted for the entire

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, Doctor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Derived] Cao X, Hu Z, Zhang Y, Wang P, Huang S, Zhu W, Dong Y, Xu H, Tang B, Zhu J. Negative-Pressure Wound Therapy Improves Take Rate of Skin Graft in Irregular, High-Mobility Areas: A Randomized Controlled Trial. Plast Reconstr Surg. 2022 Dec 1;150(6):1341-1349. doi: 10.1097/PRS.0000000000009704. Epub 2022 Sep 27. PMID 36161796